CLINICAL TRIAL: NCT00201552
Title: Atorvastatin Decreases Atrial Fibrillation Burden in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Statin and PAF in Patients With Pacemaker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 930106
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

INTERVENTIONS:
Drug: Statin

SUMMARY:
Statin could decrease AF burden

DETAILED DESCRIPTION:
Statin could decrease AF burden in patients with PAF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pacemaker

Exclusion Criteria:

* Patients with hepatic dysfunction

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jiunn-Lee Lin, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan